CLINICAL TRIAL: NCT05870267
Title: Biomechanical Assessment of Load Applied on Residuum of Individuals With Limb Loss Fitted With a Prosthetic Limb
Status: Recruiting | Type: Observational
Sponsor: YourResearchProject Pty Ltd (Industry)
Collaborators: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-YRP-LLA-Load-01
Record Dates: First submitted 2021-09-09; First posted 2023-05-23 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Prosthesis User; Amputation
Keywords: Artificial Limbs; Bone-anchored prosthesis; Bionics; Kinetics; Loading

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cohort 1 (arms 1-3): * Arm 1 will be designed as observational study providing the efficacy and safety of the load applied on osseointegrated fixation by transfemoral BAP fitted with the Power Knee for the whole cohort of 20 participants.
  * Arm 2 will be designed as matched case-control study comparing the efficacy and safety the load applied on osseointegrated fixation by transfemoral BAP fitted with Power Knee and usual MPKs (e.g., C-Leg, Genium) for the whole cohort of 20 participants.
  * Arm 3 will be designed as matched case-control study comparing the efficacy and safety the load applied on osseointegrated fixation by transfemoral BAP fitted with Power Knee and Rheo Knee XC for a subgroup of 5 participants.
  Interventions: Device: Power Knee with bone anchored suspension; Device: C-Leg; Device: Rheo Knee XC
- Cohort 2 (arm 4): • Arm 4 will be designed as matched case-control study comparing the efficacy and safety the load applied on osseointegrated fixation by transfemoral BAP fitted with Power Knee for the whole cohort of 20 participants and non-MPKs for another cohort of 10 participants.
  Interventions: Device: Power Knee with bone anchored suspension

INTERVENTIONS:
Device: Power Knee with bone anchored suspension — Motor powered microprocessor controlled prosthetic knee joint
Device: C-Leg — Passive hydraulic microprocessor controlled prosthetic knee joint
  Groups: Cohort 1 (arms 1-3)
Device: Rheo Knee XC — Passive magneto-rheologic microprocessor controlled knee joint
  Groups: Cohort 1 (arms 1-3)

SUMMARY:
This study will aim at performing biomechanical analyses of the actual load applied on the end of the stump (residuum) of individuals with transfemoral limb loss fitted with bionics bone-anchored prostheses during activities of daily living. The assessment of the inner prosthetic loading will rely on the analyses of common activities of daily living (e.g., walking in straight line and around circles, ascending and descending stairs and slopes, cycling, etc.) performed in experimental and/or clinical and/or open environments.

The biomechanical analyses of the load will address the following research questions:

A. What is the actual magnitude of the forces and moments applied on transfemoral osseointegrated implant by Rheo Knee and Power Knee during activities of daily living? living? B. What are the determinants of the loading profile in relation to the demographic and anthropometric characteristics, the type and level of activities as well as type, fitting and alignment of Rheo Knee and Power Knee? C. How the loading profiles applied by Rheo Knee and Power Knee compared to usual MPKs and Non-MPK considered below standard of care?

Biomechanical data will be collected through a typical cross-sectional cohort study. Each participant will be assessed with a given prosthesis at one particular time (i.e., exposure and outcomes will be both measured at the same time). These biomechanical analyses will rely on already published protocols (e.g., study design, instrumentation setup, extraction of loading profile). Protocols to record load data have been well described by PI-Frossard in over 20 peer-review publications in top-ranked journals. The protocol used in this study has been acknowledged, validated and are commonly used within the fields of biomechanics and prosthetics.

The outcome of this study will increase the basic understanding about the effects of loading on the interaction between body and prosthesis (e.g., osseointegration between residual bone and implant). The study will also increase applied knowledge required to establish stronger evidence-based rehabilitation programs, fitting of prosthetic limbs and design of bionics prosthetic components.

It is anticipated that, both basic and applied knowledge gain in this study will, all together, contribute to increase the health-related quality of life of individuals fitted with socket and bone-anchored prostheses.

DETAILED DESCRIPTION:
Design Biomechanical data will be collected through a typical cross-sectional cohort study. Each participant will be assessed with a given prosthesis at one particular time (i.e., exposure and outcomes will be both measured at the same time).

Arms

The whole observational study will involve a total of 30 participants (20 prospective and 10 retrospective data sets) considered in the following fours arms:

* Arm 1 will be designed as observational study providing the efficacy and safety of the load applied on osseointegrated fixation by transfemoral BAP fitted with the Power Knee for the whole cohort of 20 participants.
* Arm 2 will be designed as matched case-control study comparing the efficacy and safety the load applied on osseointegrated fixation by transfemoral BAP fitted with Power Knee and usual microprocessor controlled knees (MPKs) (e.g., C-Leg, Genium) for the whole cohort of 20 participants.
* Arm 3 will be designed as matched case-control study comparing the efficacy and safety the load applied on osseointegrated fixation by transfemoral BAP fitted with Power Knee and Rheo Knee XC for a subgroup of 5 participants.
* Arm 4 will be designed as matched case-control study comparing the efficacy and safety the load applied on osseointegrated fixation by transfemoral BAP fitted with Power Knee for the whole cohort of 20 participants and non-MPKs for another cohort of 10 participants.

Only arms 1 to 3 will involve new recording of the loading profile as part of the prospective cross-sectional cohort study for a total of 20 participants. Arms 4 will constitute the retrospective part of the study.

The data collection in Arms 1 to 3 will be organised around:

* Sessions including back-to-back successive testing of participants over a few days.
* Testing including 24 tasks enabling the recording of all the data (e.g., kinetic, video, experience) for a participant fitted with three knees (e.g., Arm 1: Power Knee, Arm 2: Usual MPKs, Arm 3: Rheo Knee).
* Recording of the loading applied on implant of participants during five trials or more of standard daily activities.

Testing:

The forces and moments applied on the three axes of the residuum, commonly referred to as the "load", were measured directly using the load cell of the iPecsLab (RTC Inc, USA). The load cell will be fitted between the participant's connector attached to the percutaneous part of the osseointegrated implant and the prosthetic knee joint.

The maximum duration of the testing will be under 6:30 hrs including 3 hrs, 3 hrs and 5 hrs requiring active participation of YourResearchProject nominated representative, Certified Prosthetist Orthotist (CPO) at APC and participant for the cohort entered in Arms 1 and 2, respectively.

The maximum duration of the testing will be under 8 hrs including 4 hrs, 4 hrs and 6:40 hrs requiring active participation of YourResearchProject nominated representative, CPO at APC and participant for the cohort entered in Arm 3, respectively.

Participants A total of 30 individuals fitted with transfemoral bone anchored prosthesis (BAP) will be asked to participate in this study. Expecting 33% drop-out rate 20 participants are expected to provide data for analysis. All participants will be asked to enter Arms 1 and 2 of the study (N=20). Five of these participants will be asked to enter Arm 3 of the study (N=5).

A tentative list of inclusion and exclusion criteria is presented in Table 1. However, the final inclusion and exclusion criteria will be discussed with CPO at APC recruiting participants.

Priority will be given to individuals treated by the team at APC who are already familiar with and, possibly, current users of MPKs including Power Knee and/or Rheo Knee XC as well as Pro-Flex XC or LP feet.

No restrictions will be placed on the ethnicity or gender of potential participants.

Recruitment Potential participants will be identified by the APC. using an arm-length method of recruitment.

Prosthesis Components Participants will be fitted with an instrumented prosthesis made of load cell and state-of-the-art components including Power Knee (Arm 1), their usual MPK (Arm 2) or Rheo Knee XC (Arm 3) as well as nominated foot/ankle units (e.g., Pro-Flex XC or LP feet) and their own footwear.

Recording Timeline The 20 participants included in Arms 1 and 2 will be asked to perform recording with Power Knee and the usual MPKs. The 5 participants selected for Arm 3 will perform an additional testing with the Rheo Knee. Altogether, the study will require a total of 20 testing.

Activities The loads will be measured while participants performed five standardized daily activities consecutively including straight level walking, ascending and descending ramp and stairs.

The recording of the actual load applied on the fixation in each activity will take place in the nominated facility (e.g., APC in Alexandria).

In all cases, a high number of gait cycles will be recorded providing sufficient number of samples to warrant comprehensive analysis if needed (e.g., statistical power).

ELIGIBILITY:
Inclusion Criteria:

* be willing to participate to this project of research,
* be able to be fitted with common bionic prosthetic components (e.g., Knee, feet),
* be willing to comply with protocol,
* have a lower limb amputation more than 12 months prior testing,
* have a clearance of at least 6 cm between residuum and prosthetic joint,
* have completed rehabilitation program,
* be free of injuries on the day of the recording session,
* weigh less than 121 kg,
* be able to walk 200 meters independently,
* be between 18-80 years of age.

Exclusion Criteria:

* not be able to give informed consent,
* have bilateral amputation,
* have self-reported pain levels greater than 4 out of 10 at study outset,
* have experienced a fall within the last 8 weeks before assessment,
* have mental illness or intellectual impairment,
* have injuries involving contralateral (intact) limb,
* have major uncorrected visual deficit,
* have history of epilepsy or recurrent dizziness,
* present signs of infection 2 weeks prior testing session.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 30 individuals fitted with transfemoral BAP will be asked to participate in this study. Drop-out rate is estimated at 33%, resulting in 20 participants completing the study. All participants will be asked to enter Arms 1 and 2 of the study (N=20). Five of these participants will be asked to enter Arm 3 of the study (N=5).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Cadence | 24 months
  Strides per minute (stride/min) corresponding to the duration between two consecutive heel contacts of the prosthetic limb measured by the load cell as described above.
Magnitude of loading pattern | 24 months
  Loading extrema correspond to onset and magnitude of a point of inflection of the loading pattern of three components of force and moment occurring consistently over successive steps, measured by the load cell as described above.
Maximum moments in gait cycle | 24 months
  Loading boundaries corresponds to the minimum, maximum and absolute maximum of the three components of forces and moments across gait cycles in relevant segment regardless of the onset, respectively, measured by the load cell as described above.

SECONDARY OUTCOMES:
The variability of datasets | 24 months
  The intra-variability of a dataset for a participant and inter-variability of a dataset between participants will be characterised by percentage of variation
Factor of safety | 24 months
  Safety of a prosthesis represented by the factor of safety ((FoS = [High impact load expressed in %BW / absolute maximum load expressed in %BW measured across all activities])) and margin of safety (MoS=FoS-1).
  MoS is calculated considering loading data for similar activities as Arms 1, 2 and 3 from the literature (e.g., Taylor et al, 2001), challenging (Edward et al, 2008) and catastrophic conditions (Ivarsson et al, 2009).
Prosthesis efficacy | 24 months
  Efficacy of a prosthesis defined as the capacity to achieve bodyweight acceptance on vertical axis that is within ±10% of full bodyweight as well as attenuate impact loads on the other axes and generate propel loads, measured by the load cell as described above.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Frossard, PhD, Principal Investigator — YourResearchProject Pty Ltd
Locations (1):
- YourResearchProject Pty Ltd, Bardon, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
Plans for return of results of research to participants:
  Feedback will be provided to individual participants about their results upon request or in cases where they could possibly benefit medically or otherwise from information collected during the study. Participants will have the options to receive their own results and the overall results of the research.
  Publication plan Scientific results will be produced through typical publication outlets (e.g., books, book chapters, manuscripts, abstract, etc.) and made available from free-access depositories (e.g., ePrint, ResearchGate) where appropriate.
  Other potential uses of the data at the end of the project The broad dissemination of the outputs will be achieved through a range of mediums including individual reports, newsletters, websites detailing the research activities, annual reports and the information sessions to be held at national and international meetings.
Time Frame: Project closure processes Retention or disposal of the documents or data will be in accordance with the Queensland State Archive University Sector Retention and Disposal Schedule for research data.
Access Criteria: Where possible, an open access approach to sharing de-identified data will be taken. At the conclusion of the project, all data will be deposited in an appropriate data repository and where appropriate non-identifiable data will be made accessible with permission.